CLINICAL TRIAL: NCT06764654
Title: Randomized Clinical Study Comparing Two Guided Surgery Techniques for Free-end Implant Placement: A Multicenter Study
Brief Title: Randomized Clinical Study Comparing Two Guided Surgery Techniques for Free-end Implant Placement
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aula Dental Avanzada (Other)
Collaborators: Mozo Grau Ticare (Unknown)
Responsible Party: Principal Investigator, Jose Antonio Sánchez-Nicolás, Principal Investigator, Aula Dental Avanzada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GUIDED
Record Dates: First submitted 2025-01-02; First posted 2025-01-08 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Dental Implant; Bone Resorption
Keywords: guided suergery; dental implant; partial edentulous
MeSH Terms: conditions — Bone Resorption

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: The operator does not know what type of surgical splint to use until the very moment of the operation, just after the anesthesia is applied.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tooth supported guide (Active Comparator): Patients who will receive implant placement using a tooth supported surgical guide.
  Interventions: Procedure: Dental implant placement
- Bone and tooth supported guide (Experimental): Patients who will receive implant placement using a bone and tooth supported surgical guide.
  Interventions: Procedure: Dental implant placement

INTERVENTIONS:
Procedure: Dental implant placement — Placement of two dental implants in the jaw.

SUMMARY:
This is a randomized multicenter clinical study that compares two static guided surgery techniques in free-end partial edentulism.

The aim is to compare the accuracy obtained between dento-osseous supported and dento-mucosal supported surgical splints to place dental implants in posterior osseous ridges.

ELIGIBILITY:
Inclusion Criteria:

* Patients who present to one of the two participating clinics with a posterior edentulous area starting from the second premolar.
* Patients in whom the placement of dental implants is not contraindicated.

Exclusion Criteria:

* Patients with hypersensitivities or allergies that contraindicate the intervention.
* Presence of orofacial neurological symptoms.
* Patients treated with bisphosphonates.
* Pregnant or breastfeeding women, or women undergoing contraceptive treatment.
* Signs of infection in the surgical area.
* Need for unconventional surgical procedures (e.g., split crest, vertical regeneration, block graft).
* Lack of patient cooperation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Three-dimensional implant position deviations (measured by intraoral scan and planning software) | From enrollment to the end of surgery
  Three-dimensional deviations between the planned implant position and the actual postoperative implant position will be assessed. The deviations will be measured using an intraoral scanner (Medit i700®) and planning software (BlueSky Plan®). Units of measure: horizontal and vertical linear deviation (in millimeters), global deviation (in millimeters), and angular deviation (in degrees), evaluated at both implant entry and apex points.

SECONDARY OUTCOMES:
Three-dimensional implant position deviations (measured by CBCT and planning software) | From enrollment to the end of surgery
  Three-dimensional deviations between the planned implant position and the actual postoperative implant position will be assessed. The deviations will be measured using cone-beam computed tomography (CBCT) and planning software (BlueSky Plan®). Units of measure: horizontal and vertical linear deviation (in millimeters), global deviation (in millimeters), and angular deviation (in degrees), evaluated at both implant entry and apex points.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Clínica Dental Esteve, Alicante, Alicante
  - Clínica Dental Sánchez Nicolás, Cabezo de Torres, Murcia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lin CC, Ishikawa M, Maida T, Cheng HC, Ou KL, Nezu T, Endo K. Stereolithographic Surgical Guide with a Combination of Tooth and Bone Support: Accuracy of Guided Implant Surgery in Distal Extension Situation. J Clin Med. 2020 Mar 5;9(3):709. doi: 10.3390/jcm9030709. PMID 32151043
- [Background] Liu R, Xia R, Zhang L, Gan X, Li C, Liu Q, Chen Z, Chen Z. The influence of guide stabilizers and their application sequences on trueness and precision of surgical guides in free end situations: An in vitro analysis. Clin Oral Implants Res. 2024 Mar;35(3):294-304. doi: 10.1111/clr.14226. Epub 2023 Dec 19. PMID 38112164
- [Background] Kessler A, Le V, Folwaczny M. Influence of the tooth position, guided sleeve height, supporting length, manufacturing methods, and resin E-modulus on the in vitro accuracy of surgical implant guides in a free-end situation. Clin Oral Implants Res. 2021 Sep;32(9):1097-1104. doi: 10.1111/clr.13804. Epub 2021 Jul 17. PMID 34218450
- [Background] Shi Y, Wang J, Ma C, Shen J, Dong X, Lin D. A systematic review of the accuracy of digital surgical guides for dental implantation. Int J Implant Dent. 2023 Oct 25;9(1):38. doi: 10.1186/s40729-023-00507-w. PMID 37875645
- [Background] Younes F, Cosyn J, De Bruyckere T, Cleymaet R, Bouckaert E, Eghbali A. A randomized controlled study on the accuracy of free-handed, pilot-drill guided and fully guided implant surgery in partially edentulous patients. J Clin Periodontol. 2018 Jun;45(6):721-732. doi: 10.1111/jcpe.12897. Epub 2018 May 10. PMID 29608793
- [Background] Cho JY, Kim SB, Ryu J. The accuracy of a partially guided system using an in-office 3D-printed surgical guide for implant placement. Int J Comput Dent. 2021 Feb 26;24(1):19-27. PMID 34006060
- [Background] Raico Gallardo YN, da Silva-Olivio IRT, Mukai E, Morimoto S, Sesma N, Cordaro L. Accuracy comparison of guided surgery for dental implants according to the tissue of support: a systematic review and meta-analysis. Clin Oral Implants Res. 2017 May;28(5):602-612. doi: 10.1111/clr.12841. Epub 2016 Apr 8. PMID 27062555
- [Background] Bover-Ramos F, Vina-Almunia J, Cervera-Ballester J, Penarrocha-Diago M, Garcia-Mira B. Accuracy of Implant Placement with Computer-Guided Surgery: A Systematic Review and Meta-Analysis Comparing Cadaver, Clinical, and In Vitro Studies. Int J Oral Maxillofac Implants. 2018 January/February;33(1):101-115. doi: 10.11607/jomi.5556. Epub 2017 Jun 20. PMID 28632253